CLINICAL TRIAL: NCT01185548
Title: The Effect of Tasisulam on the CYP2C9-Mediated Metabolism of Tolbutamide: A Pharmacokinetic Interaction Study in Cancer Patients With Advanced and/or Metastatic Solid Tumors or Lymphoma
Brief Title: A Drug Interaction Study of Tasisulam in Patients With Advanced Cancer or Lymphoma
Acronym: JZAR
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated based on safety results from another trial
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13076; H8K-MC-JZAR (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-08-18; First posted 2010-08-20 (Estimated); Results first posted 2018-10-19 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-03

CONDITIONS: Lymphoma; Advanced Cancer
Keywords: Advanced or Metastatic Solid Tumors or Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Tolbutamide; N-((5-bromo-2-thienyl)sulfonyl)-2,4-dichlorobenzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tasisulam and Tolbutamide (Experimental): Three study periods and continued access to tasisulam every 28 days (except Period 1 which was tolbutamide only and lasted 4 days) until disease progression:
  Period 1: 500 milligram (mg) tolbutamide administered on Day 1.
  Period 2: 500 mg of tolbutamide and individualized tasisulam dose [based on area under the curve albumin-corrected threshold (AUCalb)]. The AUCalb is a surrogate marker for unbound tasisulam, and this dosing approach represents the maximum level of unbound tasisulam which may be achieved clinically, administered on Day 1.
  Period 3: Individualized tasisulam dose (based on AUCalb) administered on Day 1 and 500 mg tolbutamide administered on Day 4.
  Interventions: Drug: Tolbutamide; Drug: Tasisulam

INTERVENTIONS:
Drug: Tolbutamide — Administered orally
Drug: Tasisulam — Administered intravenously
  Other Names: LY573636

SUMMARY:
The purpose of this study was to assess the effect of tasisulam as an inhibitor of CYP2C9, using tolbutamide as a probe substrate. This study was to have 3 treatment periods, and continued access in an extension period. Period 1 is 4 days in length. Periods 2 and 3 are each approximately 28 days in length. Due to the early termination of the trial, only 1 Period 3 participant enrolled in the extension period before study termination.

ELIGIBILITY:
Inclusion Criteria:

1. Have histologically or cytologically confirmed solid malignancy or lymphoma that is advanced and/or metastatic disease which has not responded to standard therapy or for which no standard therapy exists.
2. Have given written informed consent prior to any study-specific procedures.
3. Have a performance status of less than or equal to 1 on the Eastern Cooperative Oncology Group (ECOG) scale and an estimated life expectancy of greater than 12 weeks.
4. Have discontinued all previous therapies for cancer, including chemotherapy, radiotherapy, cancer-related hormonal therapy, or other investigational therapy for at least 30 days (45 days for mitomycin-C or nitrosoureas) prior to study enrollment and recovered from the acute effects of therapy. Limited field radiotherapy is permitted (in consultation with the investigator).
5. Have adequate organ function.
6. Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures.
7. Males and females with reproductive potential must agree to use medically approved contraceptive precautions during the trial and for 6 months following the last dose of study drug.
8. Females with child-bearing potential must have had a negative serum pregnancy test less than 7 days prior to the first dose of study drug.

Exclusion Criteria:

1. Have received treatment within 30 days of the initial dose of study drug with an experimental agent for noncancer indications that has not received regulatory approval for any indication.
2. Have known allergies to tasisulam or related compounds.
3. Have serious preexisting medical conditions.
4. Show evidence of significant active neuropsychiatric disease or central nervous system (CNS) disease (for example, Alzheimer's disease or Parkinson's disease). Patients with active brain metastasis are excluded.
5. Have current acute or chronic leukemia.
6. Females who are pregnant or lactating.
7. Have known positive test results in human immunodeficiency virus (HIV), hepatitis B surface antigen (HBSAg), or hepatitis C antibodies (HCAb).
8. History of severe allergies or multiple adverse drug reactions.
9. Are persons who have previously completed or withdrawn from this study or any other study investigating tasisulam.
10. Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study.
11. Serious concomitant systemic disorder, including diabetes or active infection, incompatible with the study.
12. Clinically significant cardiac symptomology.
13. Patients being treated with warfarin.
14. Patients being treated with sulfonylureas
15. Regularly use drugs of abuse and/or show positive findings on urinary drug screening that is not in accordance with known/acceptable concomitant medication.
16. Patients who have received medications that are known inducers or inhibitors of CYP2C9 within 30 days prior to enrollment.
17. Have donated or lost blood of more than 500 milliliter (mL) within the last month.
18. Have an average weekly alcohol intake that exceeds 21 units per week (males up to age 65) and 14 units per week (males over 65 and females) (1 unit = 12 ounces (oz) or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits).
19. Failure for any reason to satisfy the investigator for adequate fitness to participate in the study.
20. Screening albumin levels less than 30 grams/Liter (g/L).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (5):
- United Kingdom (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cardiff, South Glamorgan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sheffield, Trent
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leeds, West Yorkshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leicester
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Period 1: 500 milligram (mg) tolbutamide administered once on Day 1
  Period 2: 500 mg of tolbutamide and individualized tasisulam dose (based on AUCalb) administered once on Day 1
  Period 3: individualized tasisulam dose (based on AUCalb) administered once on Day 1 and 500 mg tolbutamide administered once on day 4
Period: Period 1 : Tolbutamide
Arm/Group | All Participants
Started | 4
Completed | 4
Not Completed | 0
Period: Period 2: Tasisulam and Tolbutamide
Arm/Group | All Participants
Started | 4
Completed | 2
Not Completed | 2
Not completed — Sponsor Decision | 2
Period: Period 3: Tasisulam and Tolbutamide
Arm/Group | All Participants
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants were included in the analysis.
Groups:
- All Participants: Three study periods: Period 1 which was tolbutamide only and lasted 4 days and Periods 2 and 3 which had continued access to tasisulam every 28 days until disease progression:
  Period 1: 500 mg tolbutamide administered once on Day 1.
  Period 2: 500 mg of tolbutamide and individualized tasisulam dose administered once on Day 1.
  Period 3: individualized tasisulam dose administered once on Day 1 and 500 mg tolbutamide administered once on Day 4.
Arm/Group | All Participants
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 4

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics of Tolbutamide, Concurrent Dosing, Area Under the Curve (AUC 0-∞)
Description: AUC0-∞ is defined as the area under the concentration time curve from time 0 to infinity.
Time Frame: Period 2 Predose; and 0.5, 1, 1.5, 2, 2.5, 3, 4, 4.5, 6, 8, 24, 48, 72, 120, 168, 336 hours post tolbutamide dose
Population: All enrolled participants who started Period 2 (tasisulam and tolbutamide).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour per milliliter (ng*hr/mL)
Groups:
- Period 2: Tasisulam and Tolbutamide: Period 2: 500 mg of tolbutamide and individualized tasisulam dose (based on AUCalb) administered once on Day 1
Arm/Group | Period 2: Tasisulam and Tolbutamide
Number analyzed (Participants) | 4
nanograms*hour per milliliter (ng*hr/mL) | 2670000 (20)

2. Secondary Outcome: Pharmacokinetics of Tolbutamide, Staggered Dosing in Period 3, Area Under the Curve (AUC 0-∞)
Description: AUC0-∞ is defined as the area under the concentration time curve from time 0 to infinity.
Time Frame: Period 3 Predose; and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 24, 48, 96, and 264 hours post tolbutamide dose
Population: All enrolled participants who started period 3 (tasisulam then tolbutamide).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Groups:
- Tasisulam and Tolbutamide: Period 3: Period 3: Individualized tasisulam dose (based on AUCalb) administered once on Day 1 and 500 mg tolbutamide administered once on Day 4.
Arm/Group | Tasisulam and Tolbutamide: Period 3
Number analyzed (Participants) | 2
nanogram*hour per milliliter (ng*hr/mL) | 2700000 (NA) [4.03 to 6] — There were not a sufficient number of participants to calculate the geometric coefficient of variation.

3. Secondary Outcome: Pharmacokinetics of Tolbutamide, Maximum Concentration (Cmax)
Time Frame: Period 1, 2, and 3 Predose; and 0.5, 1, 1.5, 2, 2.5, 3, 4, 4.5, 6, 8, 24, 48, 72, 96, 120, 168, 264, 336 hours post tolbutamide dose
Population: All enrolled participants who started Periods 1, 2, or 3.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- Tolbutamide: Period 1: Period 1: 500 mg tolbutamide administered once on Day 1
- Tasisulam and Tolbutamide: Period 2: Period 2: 500 mg of tolbutamide and individualized tasisulam dose (based on AUCalb) administered once on Day 1.
Arm/Group | Tolbutamide: Period 1 | Tasisulam and Tolbutamide: Period 2 | Tasisulam and Tolbutamide: Period 3
Number analyzed (Participants) | 4 | 4 | 2
nanogram per milliliter (ng/mL) | 39600 (26) | 39800 (18) | 48000 (NA) — There were not a sufficient number of participants to calculate the geometric coefficient of variation.

4. Secondary Outcome: Pharmacokinetics of Tolbutamide, Observed Time at Maximal Concentration (Tmax)
Time Frame: as for outcome 3
Population: All enrolled participants who started Periods 1, 2, or 3.
Measure: Median (Full Range); unit: hours
Groups:
- Period 1: Tolbutamide: Period 1: 500 mg tolbutamide administered once on Day 1
- Period 2: Tasisulam and Tolbutamide: Period 2: 500 mg tolbutamide and an individualized tasisulam dose (based on AUCalb) administered once on Day 1.
- Period 3: Tasisulam and Tolbutamide: Period 3: Individualized tasisulam dose (based on AUCalb) administered once on Day 1 and 500 mg tolbutamide administered once on day 4 (administration day in period 3 could adjusted based on interim pharmacokinetic [PK] analyses)
Arm/Group | Period 1: Tolbutamide | Period 2: Tasisulam and Tolbutamide | Period 3: Tasisulam and Tolbutamide
Number analyzed (Participants) | 4 | 4 | 2
hours | 2.25 [2.00 to 3.00] | 5.00 [1.50 to 8.00] | 5.02 [4.03 to 6.00]

ADVERSE EVENTS:
Groups:
- Tolbutamide: Adverse events (AEs) that occurred during Period 1 and during Period 2 when 500 mg tolbutamide was administered orally prior to individualized intravenous dosing (based on AUCalb) of tasisulam.
- Tasisulam and Tolbutamide: AEs that occurred during Periods 2 and 3 when both 500 mg oral tolbutamide and individualized intravenous tasisulam (based on AUCalb) were administered.
- Tasisulam: AEs that occurred during Period 3 Day 1 through Day 4 until just before 500 mg oral tolbutamide was administered on Day 4, 72 hours.
Arm/Group | Tolbutamide | Tasisulam and Tolbutamide | Tasisulam
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/4 | 0/2
Other Adverse Events (participants affected / at risk) | 3/4 | 4/4 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tolbutamide (N=4) | Tasisulam and Tolbutamide (N=4) | Tasisulam (N=2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tolbutamide (N=4) | Tasisulam and Tolbutamide (N=4) | Tasisulam (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (4) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Jessner's lymphocytic infiltration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days